CLINICAL TRIAL: NCT00855816
Title: PTSD Hyperarousal Symptoms Treated With Physiological Stress Management
Brief Title: Post Traumatic Stress Disorder (PTSD) Hyperarousal Symptoms Treated With Physiological Stress Management
Acronym: BaRT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MHBA-019-08F
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Breathing training (Experimental): relaxation training
  Interventions: Behavioral: Breathing training
- Treatment as usual (No Intervention): treatment as usual

INTERVENTIONS:
Behavioral: Breathing training — relaxation training
  Arms: Breathing training

SUMMARY:
Hyperarousal is a key symptom of PTSD. Even after receiving trauma-focused therapy, PTSD patients may continue to suffer from hyperarousal. Our main objectives are to measure hyperarousal in VA outpatients with PTSD related to combat experience in the last 10 years and to test the efficacy of physiological relaxation training in reducing this hyperarousal. Measurements will be both physiological, using 24 hour ambulatory monitoring of skin conductance, heart rate, and physical activity during waking and sleeping, and psychological, using self-reports and clinician interviews. Specific aims include initially evaluating 100 or more PTSD patients for the severity of their hyperarousal symptoms. Of these, 50 with at least moderate hyperarousal who either have participated in a trauma-focused therapy or have declined to participate in such a therapy will be recruited for a therapy trial. Volunteers will be randomized to treatment consisting of 5 sessions of individual physiological relaxation training with biofeedback over a 4-week period or to a 2-month waiting period after which they also may receive this therapy. Physiological evaluations of the patients' ability to relax will be measured at three times -before treatment, immediately after treatment, and 6 months after treatment. Clinical evaluations by interviews and questionnaires on measures of symptoms and disability will be measured at four times - before treatment, immediately after treatment, 1 month after treatment, and 6 months after treatment. The waiting-list group and a nonanxious control group will be tested psychophysiologically twice at the same interval as the patients before and immediately after treatment. A control group will allow us to calibrate our measures in the setting in which they are being applied. We hypothesize that this therapy will relieve both self-reported and objective, physiological symptoms of hyperarousal.

Relevance to health and the VA mission: Many of our clients at the VA Palo Alto Mental Health Outpatient Services for PTSD are veterans of Iraq, who need help with hyperarousal symptoms. This study will fill in gaps in our knowledge about the physiology of these symptoms and about the efficacy of relaxation therapies. Non-pharmacological treatments like the ones that we propose may relieve patients' hyperarousal to an extent that they are less tempted to turn to alcohol or sedative drugs.

DETAILED DESCRIPTION:
Hyperarousal is a key symptom of PTSD. Even after receiving trauma-focused therapy, PTSD patients may continue to suffer from hyperarousal. Neuroimaging findings in PTSD support the idea that regulation of autonomic arousal from the cingulate cortex can be helpful in reducing anxiety.

Our main objectives are to measure hyperarousal in VA outpatients with PTSD related to combat experience in the last 10 years and to test the efficacy of physiological relaxation training in reducing this hyperarousal. Measurements will be both physiological, using 24 hour ambulatory monitoring of skin conductance, heart rate, and physical activity during waking and sleeping, and psychological, using self-reports and clinician interviews. Specific aims include initially evaluating 100 or more PTSD patients for the severity of their hyperarousal symptoms. Of these, 50 with at least moderate hyperarousal who either have participated in a trauma-focused therapy or have declined to participate in such a therapy will be recruited for a therapy trial. Volunteers will be randomized to treatment consisting of 5 sessions of individual physiological relaxation training with electromyographic feedback and with capnographic feedback over a 4-week period or to a 2-month waiting period after which they also may receive this therapy. Physiological evaluations of the patients' ability to relax while sitting quietly and their arousal levels during daily activities and sleep will be measured at three times -before treatment, immediately after treatment, and 6 months after treatment. Clinical evaluations by interviews and questionnaires on measures of symptoms and disability will be measured at four times - before treatment, immediately after treatment, 1 month after treatment, and 6 months after treatment. The waiting-list group and a nonanxious control group will be tested psychophysiologically twice at the same interval as the patients before and immediately after treatment. A control group will allow us to calibrate our measures in the setting in which they are being applied. We hypothesize that this therapy will relieve both self-reported and objective, physiological symptoms of hyperarousal.

Relevance to health and the VA mission: Many of our clients at the VA Palo Alto Mental Health Outpatient Services for PTSD are veterans of Iraq, who need help with hyperarousal symptoms. This study will fill in gaps in our knowledge about the physiology of these symptoms and about the efficacy of relaxation therapies. Non-pharmacological treatments like the ones that we propose may relieve patients' hyperarousal to an extent that they are less tempted to turn to alcohol or sedative drugs. Physiological proof of the effectiveness of relaxation procedures in this clinical group would help convince clinicians to apply them and patient consumers to try them.

ELIGIBILITY:
Inclusion Criteria:

*Participants in the PTSD treatment MUST be US military veterans. Healthy volunteers may include members of the general community, as well as veterans or active duty military personnel*

* Patients diagnosed by DSM-IV criteria for current PTSD,
* OR met DSM-IV criteria for PTSD within last 5 years.
* Patients must either have participated in a trauma-focused therapy,
* OR have declined to participate in such a therapy.
* In addition, they must currently score positive on at least 2 of the 5 D criteria symptoms.

This will be defined as having a CAPS frequency plus intensity ratings greater than or equal to 4.

Exclusion Criteria:

* Patients with evidence of current significant alcohol abuse or dependence, psychosis, or substantial cognitive deficits,
* OR who are severely depressed or acutely suicidal and will not be accepted until these problems are resolved.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-02; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walton Roth, MD, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

REFERENCES:
- [Derived] Jamison AL, Slightam C, Bertram F, Kim S, Roth WT. Randomized clinical trial of capnometry-assisted respiratory training in veterans with posttraumatic stress disorder hyperarousal. Psychol Trauma. 2022 Jul;14(5):883-893. doi: 10.1037/tra0000525. Epub 2019 Dec 5. PMID 31804108
- [Derived] Slightam C, Petrowski K, Jamison AL, Keller M, Bertram F, Kim S, Roth WT. Assessing sleep quality using self-report and actigraphy in PTSD. J Sleep Res. 2018 Jun;27(3):e12632. doi: 10.1111/jsr.12632. Epub 2017 Nov 24. PMID 29171107

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment as Usual: No intervention - treatment as usual
Period: Overall Study
Arm/Group | Breathing Training | Treatment as Usual
Started | 47 | 33
Completed | 21 | 12
Not Completed | 26 | 21
Not completed — Withdrawal by Subject | 22 | 15
Not completed — Lost to Follow-up | 3 | 5
Not completed — Death | 1 | 0
Not completed — Became ineligible | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment as Usual: No intervention: Treatment as usual
- Total: Total of all reporting groups
Arm/Group | Breathing Training | Treatment as Usual | Total
Number analyzed (Participants) | 47 | 33 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.09 (11.04) | 53.21 (10.62) | 53.14 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 40 | 30 | 70
Region of Enrollment [Number; unit: participants]
  United States | 47 | 33 | 80

OUTCOME MEASURES:

1. Primary Outcome: Change Scores for Criteria D Items on the CAPS Structured Clinical Interview
Description: Change in total score for all criterion D items on the Clinician-Administered PTSD Scale for DSM-IV, from baseline to post-treatment.
  Total Criterion D subscore = sum of all frequency (0-4) and intensity (0-4) ratings of 5 PTSD hyperarousal symptoms.
  Range: 0 to 40, with higher scores indicating more severe (frequent and/or intense) symptoms.
  Change score calculated as: CAPS D score time 2 - CAPS D score time 1. Greater negative change scores indicate greater reduction in symptom severity (aka symptom improvement).
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Breathing Training | Treatment as Usual
Number analyzed (Participants) | 47 | 33
units on a scale | -1.20 (4.41) | -6.27 (6.22)
Statistical Analysis 1: Comparison: Breathing Training vs Treatment as Usual; Null hypothesis: there will be no differences in PTSD hyperarousal symptom changes in individuals who did receive the experimental intervention vs. those who did not; Test type: Superiority or Other; p = .27, Mixed Models Analysis — A priori threshold for significance: p<.05; Mixed model based on intent to treat sample

ADVERSE EVENTS:
Arm/Group | Breathing Training | Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 3/47 | 1/33
Other Adverse Events (participants affected / at risk) | 0/47 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Breathing Training (N=47) | Treatment as Usual (N=33)
Hospitalization (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — Unplanned knee surgery
Death (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Multiple myeloma
Hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) — Alcohol and drug relapse

LIMITATIONS AND CAVEATS:
Higher than anticipated withdrawal rate limited power of statistical analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No